CLINICAL TRIAL: NCT00537563
Title: AMS VS MOXI Ketek vs Avelox in AMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMR3647A_4017
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Maxillary Sinusitis
MeSH Terms: conditions — Maxillary Sinusitis | interventions — telithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Telithromycin

SUMMARY:
Clinical efficacy between telithromycin and moxifloxacin at the post-therapy/test of cure visit, and to assess the safety of telithromycin given once daily for 5 days vs moxifloxacin given once daily for 10 days in the treatment of subjects with AMS.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects, aged 18 years or older, AMS diagnosed (clinically and radiologically) who were willing to undergo rhinoscopic aspiration or deep nasal swab at the baseline/pre-therapy visit. Female subjects of childbearing potential were required to have a negative pregnancy test before undergoing any study procedure and to use an accepted contraceptive method during the study.

Exclusion Criteria:

* Women who were breast-feeding or pregnant, as demonstrated by serum or urine pregnancy tests carried out before exposure to study medication or the start of any study procedure that could pose a risk to the fetus;
* Subjects with a history of recurrent sinusitis (defined as more than 3 episodes of sinusitis that required antibiotic therapy in the preceding 12 months);
* Subjects with a history of chronic sinusitis (defined as symptoms lasting greater than 28 days);
* Subjects with sphenoidal sinusitis involvement that required treatment other than oral antibiotics;
* Subjects with nosocomial-acquired sinusitis within 2 weeks (eg, hospitalization or nonambulatory, institutional confinement, including nursing homes);
* Subjects with any concomitant medication [including functionally significant, major obstructive anatomical lesions likely to impair resolution of infection (eg, nasal polyps extending past the middle turbinate, tumor, or severe septal deviation)], such as: asthma, cystic fibrosis, immotile cilia syndrome, prior nasopharyngeal or sinus surgery, sinus polyps, clinically relevant cardiovascular (eg, congestive heart failure), neurologic, endocrine, or other major systemic disease that could have made implementation of the protocol or interpretation of the study results difficult;
* Subjects with a need for immediate surgery for maxillary sinusitis;
* Subjects who used nasal, nasogastric, or nasotracheal catheters;
* Subjects with previous sinus surgery within the past 6 months or sinus lavage within the past 7 days;
* Subject who were long-term (> than or = to 4 weeks) users of nasal decongestants like oxymetazoline 0.05%;
* Subjects with suspected nonbacterial infections;
* Subjects with a concomitant odontological infection that would require antibiotic therapy or surgery;
* Subjects with unknown or suspected hypersensitivity to, or a known or suspected serious adverse reaction to either study medication, any fluoroquinolone, or any macrolide antibiotic;
* Subjects who would likely have required on-study treatment with drugs known to have contraindicated drug interactions with either study medication and/or macrolides or fluoroquinolones in general, including, but not limited to: ergot alkaloid derivatives, cholinesterase inhibitors (eg, tacrine, donepezil, physostigmine) ketamine, carbamazepine, St John's Wort, Class IA (eg, quinidine, procainamide), or Class III antiarrhythmic agents (eg, amiodarone, sotalol);
* Subjects who required anticoagulant therapy (eg, warfarin);
* Subjects who received treatment with other systemic antibiotics (oral or parenteral) within 14 days prior to study enrollment;
* Subject who received moxifloxacin or another fluoroquinolone antibiotic for this infectious episode;
* Likelihood of required treatment during the study period with drugs not permitted by the protocol;
* Treatment with any investigational product in the last 1 month prior to study entry;
* Subjects with a progressively fatal disease; life expectancy <less than or = to 3 months;
* Clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult;
* History of drug or alcohol abuse;
* Impaired hepatic function [as shown by previous clinical laboratory values of AST (SGOT) and/or ALT (SGPT) > than or = to 3 times the upper limit of reference range, total bilirubin > than 2 times the upper limit of reference range (except for Gilbert's disease), encephalopathy, etc];
* Impaired renal function [as shown by previous clinical laboratory values of creatinine clearance < than or = to 30 mL/min (< than or = to 0.50 mL/sec), serum creatinine > than or = to 2.0 mg/dl (> than or = to 176 micromol/L), etc]. Creatinine clearance may have been estimated by formula or by nomogram;
* Immunocompromised subjects, such as subjects with HIV infection and who had either an AIDS-defining condition (eg, Kaposi's sarcoma and Pneumocystis carinii pneumonia), or a CD4 + T-lymphocyte count of < 200/mm3). A complete list is provided in Appendix 3 of the clinical study protocol (see @@Appendix A.1.1).
* subjects with neutropenia (<1500 neutrophils/mm3) not attributable to the acute infectious disease
* subjects with metastatic or hematological malignancy
* splenectomised subjects with known hyposplenia or asplenia
* subjects with known IgG deficiency
* Subject with known long QT syndrome or familiar history of long QT syndrome (if no previous ECG has invalidated this risk factor), or personal history of coronary disease, ventricular arrhythmia, bradycardia < 50 beats/min, or known uncorrected hypokalemia or hypomagnesemia, or who were treated with concomitant medication known to prolong QT interval (eg, cisapride, pimozide, astemizaole, terfenadine, or potent CYP3A4 inhibitors, such as: protease inhibitors, ketoconazole);
* Mental condition that rendered the subject unable to understand the nature, scope, and possible consequences of the study;
* Subjects diagnosed with myasthenia gravis (ie, Protocol Amendment No. 1);
* Subjects unlikely to comply with the protocol (eg, uncooperative attitude, inability to return for follow-up visit, and unlikely to complete the study);
* Subjects without a permanent residential address or home telephone number;
* Any waiver of these inclusion/exclusion criteria was to be approved by the investigator and Aventis on a case-by-case basis, prior to study enrollment. This was to be documented by both the investigator and Aventis; or
* No subject was allowed to enroll in this study more than once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2002-12; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
To demonstrate equivalence in clinical efficacy between telithromycin and moxifloxacin at the post-therapy/test of cure (TOC) visit. | Days 17 to 24

SECONDARY OUTCOMES:
Assess the safety of telithromycin given once daily for 5 days vs moxifloxacin given once daily for 10 days in the treatment of subjects with AMS.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States